CLINICAL TRIAL: NCT00912873
Title: Optimizing Local Anesthetic Concentration for Continuous Lumbar Plexus Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hip Concentration Study
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Hip Arthroplasty; Hip Pain
Keywords: postoperative pain; perineural catheter; continuous peripheral nerve block; posterior lumbar plexus; hip surgery; psoas compartment; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.1% Ropivicaine (Active Comparator): Patients will be given 0.1% ropivicaine provided via infusion pump which will be attached intraoperatively and will remain connected until patient is ready to leave the hospital. In this time a physical therapist will work with the patient to assess outcome measures.
  Interventions: Drug: 0.1% Ropivacaine
- 0.4% Ropivicaine (Experimental): Patients will be given 0.4% ropivicaine provided via infusion pump which will be attached intraoperatively and will remain connected until patient is ready to leave the hospital. In this time a physical therapist will work with the patient to assess outcome measures.
  Interventions: Drug: 0.4% Ropivacaine

INTERVENTIONS:
Drug: 0.1% Ropivacaine — Ropivacaine 0.1% will be administered via the perineural catheter as follows: Basal Rate (12mL/h); Basal Dose (12 mg/h); Bolus Volume (4 mL); Bolus Dose (4 mg); Lockout Duration (30 min); Maximum Dose (20 mg/h)
  Arms: 0.1% Ropivicaine
Drug: 0.4% Ropivacaine — Ropivacaine 0.1% will be administered via the perineural catheter as follows: Basal Rate (3 mL/h); Basal Dose (12 mg/h); Bolus Volume (1 mL); Bolus Dose (4 mg); Lockout Duration (30 min); Maximum Dose (20 mg/h)
  Arms: 0.4% Ropivicaine

SUMMARY:
This is a research study to determine if the concentration of local anesthetic through a catheter next to the nerves that go to the hip that is undergoing surgery, affects muscle strength and sense of touch experienced after surgery. This study is looking at the varying concentrations of local anesthetic placed through the catheter.

DETAILED DESCRIPTION:
These results will help define the optimal concentration of local anesthetic used for continuous peripheral nerve blocks and help guide future research in this clinically-relevant area.

This investigation will be a randomized, observer-masked, controlled, parallel-arm, human-subjects clinical trial.

Enrollment. Subjects will be patients undergoing hip arthroplasty. Study inclusion will be proposed to eligible patients by the orthopedic surgery or anesthesia services or research coordinator/assistant within four weeks prior to surgery. If a patient desires study participation, written, informed consent will be obtained. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status.

Preoperative Management. Prior to surgery but following written, informed consent, subjects will have baseline endpoints measured. Patients will then have a perineural catheter placed on the operative side using standard techniques currently used at UCSD, and previously described. A 15 mL bolus of 2% mepivacaine with epinephrine (5 µg/mL) will be injected through the catheter to demonstrate correct catheter placement and provide intraoperative analgesia. Patients with a misplaced catheter indicated by a lack of sensory changes in the surgical extremity within 15 min will have their catheter replaced or be withdrawn from the study prior to randomization.

The remaining patients will then be randomized to one of two treatment groups: a postoperative ropivacaine concentration of 0.1% or 0.4% ("study infusate"). Randomization will be based on computer-generated codes that will be created and maintained by the Investigational Drug Service. Randomization will be in blocks of four, and stratified by hip arthroplasty procedure (either total or resurfacing). A portable electronic infusion pump with study infusate will be attached to the perineural catheter. The basal rate and patient-controlled bolus volume will depend upon the treatment group (note that the basal rate and bolus volume differ for each concentration, but the total dose of local anesthetic is the same for each):

Ropivacaine Concentration 0.1%: Basal Rate (12mL/h); Basal Dose (12 mg/h); Bolus Volume (4 mL); Bolus Dose (4 mg); Lockout Duration (30 min); Maximum Dose (20 mg/h)

Ropivacaine Concentration 0.4%: Basal Rate (3 mL/h); Basal Dose (12 mg/h); Bolus Volume (1 mL); Bolus Dose (4 mg); Lockout Duration (30 min); Maximum Dose (20 mg/h)

Intraoperative Management. Patients will receive a standardized general anesthetic with an inhaled anesthetic in N2O and O2. These gasses will be titrated for a Bispectral Index of 40-60 in order to provide adequate anesthesia while minimizing postoperative recovery duration. Esmolol and hydralazine will be used to provide hemodynamic stability, and opioids administered if necessary (fentanyl in 25 µg increments). The ropivacaine infusion provided by the Investigational Drug Service will be initiated using an infusion pump attached to the perineural catheter. Just prior to emergence, IV morphine will be titrated for a respiratory rate of 12-14. Upon emergence, patients will be taken to the recovery room and then to the surgical ward.

Postoperative Pain Management. For the duration of the study, all patients will receive the current usual and customary analgesics for hip arthroplasty patients at Hillcrest and Thornton hospitals. Perineural infusions will be administered per standard UCSD routine: continued administration until recommended discontinuation by the surgical service at which time the catheter is removed by the acute pain service.

Outcome Measurements. We have selected measures that have established reliability and validity. Staff blinded to treatment group assignment will perform all measures and assessments. Preoperative measurements (performed prior to perineural catheter placement the day of surgery): strength of the quadriceps femoris, hip adductors, and hip flexors; and sensory level (measurement descriptions below). Postoperative measurements will be performed the day following surgery as close to 8:00-9:00 and 12:30-13:30 as possible (logistics occasionally preclude therapist evaluation at these exact hours).

ELIGIBILITY:
Inclusion Criteria:

* Primary, unilateral hip arthroplasty
* age greater than or equal to 18 years
* postoperative analgesic plan includes perineural local anesthetic infusion

Exclusion Criteria:

* morbid obesity as defined by a body mass index greater than 40
* chronic high dose opioid use
* history of opioid abuse
* neuro-muscular deficit of the ipsilateral femoral nerve and/or quadriceps muscle
* vulnerable populations i.e., children, pregnant women, or prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilfeld BM, Moeller LK, Mariano ER, Loland VJ, Stevens-Lapsley JE, Fleisher AS, Girard PJ, Donohue MC, Ferguson EJ, Ball ST. Continuous peripheral nerve blocks: is local anesthetic dose the only factor, or do concentration and volume influence infusion effects as well? Anesthesiology. 2010 Feb;112(2):347-54. doi: 10.1097/ALN.0b013e3181ca4e5d. PMID 20098137

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.1% Ropivicaine: ropivicaine 0.1% infusion at 12 mL/hour
- 0.4% Ropivicaine: ropivicaine 0.4% infusion at 3 mL/hour
Period: Overall Study
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.1% Ropivicaine: ropivicaine 0.1% infusion at 3 mL/hour
- Total: Total of all reporting groups
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (3) | 52 (4) | 52.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 15 | 15 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Quadriceps Femoris Maximum Voluntary Isometric Contraction (MVIC)
Description: Quadriceps femoris muscle strength evaluated using a portable, hand-held, isometric force dynamometer (MicroFET2, Lafayette Instrument Company, Lafayette, IN) to measure the maximum voluntary isometric contraction (MVIC) in a seated position. The study primary endpoint will be the difference in MVIC the morning following surgery compared with the preoperative MVIC, expressed as a percentage of the preoperative MVIC: (preop - postop ) / preop x 100.
Time Frame: The study primary endpoint will be the difference in MVIC the morning following surgery compared with the preoperative MVIC, expressed as a percentage of the preoperative MVIC: (preop - postop ) / preop x 100.
Measure: Mean (Standard Error); unit: percentage change from baseline of MVIC
Groups:
- 0.1% Ropivicaine: 0.1% Ropivicaine at 12 mL/h
- 0.4% Ropivicaine: 0.4% Ropivicaine at 3 mL/h
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
percentage change from baseline of MVIC | 64.1 (6.4) | 68 (5.4)

2. Secondary Outcome: Ambulation 100-foot Walking Test
Description: The 100-foot walking test simply measures the amount of time it takes patients to ambulate 100 feet. Patients will be allowed to slow or stop and rest during the walk, but will be asked to resume walking as soon as they feel they are able to.
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: minutes
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
minutes
  Morning | 4.6 (0.3) | 5.3 (0.2)
  Afternoon | 4.0 (0.3) | 3.6 (0.3)

3. Secondary Outcome: Total Ambulation
Description: Patients will be allowed to slow or stop and rest during the walk, but will be asked to resume walking as soon as they feel they are able to and go as far as they comfortable walking.
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: meters
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
meters
  morning | 136 (23) | 119 (16)
  afternoon | 223 (43) | 214 (36)

4. Secondary Outcome: Percent Change From Baseline in Hip Flexion
Description: Evaluated in the supine position using a portable, hand-held, isometric force dynamometer (MicroFET2, Lafayette Instrument Company, Lafayette, IN). The endpoint will be the difference the morning following surgery compared with the preoperative value, expressed as a percentage of the preoperative value: (preop - postop ) / preop x 100.
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: percentage change from baseline hip flex
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
percentage change from baseline hip flex
  morning | 69 (4) | 67 (3)
  afternoon | 75 (3) | 78 (36)

5. Secondary Outcome: Mean Resting Pain
Description: Pain level evaluated using a verbal rating scale of 0-10, with 0=no pain and 10=worst imaginable pain
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
units on a scale | 3.2 (0.4) | 3.2 (0.4)

6. Secondary Outcome: Average Dynamic Pain
Description: Pain evaluated during physical therapy using a verbal rating scale of 0-10, with 0=no pain and 10=worst imaginable pain
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
units on a scale
  morning | 3.8 (0.4) | 3.8 (0.4)
  afternoon | 3.2 (0.4) | 2.9 (0.3)

7. Secondary Outcome: Worst Dynamic Pain
Description: The worst pain experienced during physical therapy evaluated using a verbal rating scale of 0-10, with 0=no pain and 10=worst imaginable pain
Time Frame: Day following surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
Number analyzed (Participants) | 26 | 24
score on a scale
  morning | 6.2 (0.5) | 6.5 (0.5)
  afternoon | 4.3 (0.4) | 5.0 (0.6)

ADVERSE EVENTS:
Time Frame: Through the day following surgery
Arm/Group | 0.1% Ropivicaine | 0.4% Ropivicaine
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No